CLINICAL TRIAL: NCT01450514
Title: POC Study of Pipamperone 15mg Added to Stable Risperidone or Paliperidone Treatment in Chronic Schizophrenic and Schizoaffective Patients With Residual Symptoms: a Phase I/IIa, Randomized, Double-blind, Placebo-controlled Trial of 7 Weeks
Brief Title: POC Study of Pipamperone Added to Stable Treatment With RIS or PAL in Chronic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaNeuroBoost N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNB02-C201; 2011-004494-81 (EudraCT Number)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Psychotic Disorders | interventions — pipamperone; Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo
- Pipamperone (Experimental): 15 mg once daily
  Interventions: Drug: Pipamperone

INTERVENTIONS:
Drug: Pipamperone — 15 mg PIP once daily per os on top of continued stable treatment with RIS or PAL
  Other Names: Risperdal, Invega and Xeplion
  Arms: Pipamperone
Drug: Placebo — matching placebo sugar pill once daily per os on top of continued stable treatment with RIS or PAL
  Arms: Placebo

SUMMARY:
This Phase I/IIa Proof-of-Concept (PoC) trial is designed to assess the effect of adding a single and repeated low dose (15mg/d) of pipamperone (PIP) for 6 weeks to stable treatment with an effective dose of risperidone (RIS) or paliperidone (PAL) on functional MRI tests and clinical outcome of chronic schizophrenic patients with residual, so-called 'positive' symptoms, as well as on cognition, motivation, subjective well-being of patients, negative symptoms, general psychopathological symptoms and safety/tolerability.

DETAILED DESCRIPTION:
This exploratory study of 7 weeks was intended to be performed in 40 to 60 patients in up to 10 centers in Belgium. In a subset of patients, the 6-week treatment phase will be preceded by a single-dose cross-over phase with 1 week of wash-out. While the objective of the study, due to its exploratory design, is to assess any effect of the study medication on MRI or clinical outcome, the study medication is expected to improve the residual (remaining) positive symptom(s) of patients. In addition, genetic and pharmacokinetic testing may be performed to learn more about the disorder and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
* Patient understands the investigational nature of the trial and is willing and able to comply with the trial requirements.
* Patient is male or female, aged 18-65 years.
* Patients has Schizophrenia or Schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV-R criteria. Diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Patient is being treated during at least 12 weeks with a stable dosage of either risperidone depot of 12.5-50mg IM every 2 weeks, paliperidone depot of 25-100mg IM every 4 weeks, risperidone oral administration of 2-6 mg/d, or paliperidone oral administration of 4-12 mg/d
* Patient has a CGI-S score of 3 (mildly ill) or more at baseline.
* Patient has a score of 4 or more on at least 1 item of the positive PANSS subscale (residual symptoms).

Exclusion Criteria:

* Acute exacerbation of schizophrenic or schizoaffective disorder during the past 12 weeks.
* Documented debility or an IQ below 85.
* Comorbid axis 1 conditions (including anxiety disorders, eating disorders, impulse control disorders) requiring drug treatment over the previous 12 weeks.
* Patient has taken, in the past 6 weeks prior to randomization, any newly initiated psychoactive drug.
* Patient was withdrawn from psychoactive drug treatment in the past week or within a period shorter than 5x the elimination half-life of any psychoactive drug. Withdrawal of any prior antipsychotic treatment should not have occurred within 6 weeks prior to baseline.
* Concomitant treatment with any additional antipsychotic drug at a therapeutic dosage, diuretics, QT prolongation drugs, or dopamine agonists.
* Formal cognitive psychotherapy initiated during study treatment or within 6 weeks prior to randomization.
* Patient has any other medical or psychiatric condition, which in the opinion of the investigator, can jeopardize or would compromise the patient's ability to participate in this trial or that would interfere with trial assessments.
* Patient with a DSM-IV alcohol or substance dependence diagnosis (within the last 6 months), an alcohol or substance abuse diagnosis (within the last month) or having a positive standard screen for alcohol or drugs (including benzodiazepines and opioids).
* 'Any concomitant psychoactive treatment (including psychotherapy)' or 'Patient received, in the 6 weeks prior to randomization any newly prescribed psychoactive drug'.
* Patient is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, 2 years postmenopausal, or who does not consistently use 2 combined effective methods of contraception (including at least 1 barrier method), unless sexually abstinent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional MRI tests | 1 day, 2 weeks and 6 weeks after study treatment start
  MRI = Magnetic Resonance Imaging Functional tests performed during MRI include the N-Back Test and the Monetary Incentive Delay (MID) Task Test

SECONDARY OUTCOMES:
Change from baseline in residual PANSS item(s) | 2 weeks and 6 weeks after study treatment start
  PANSS = Positive and Negative Syndrome Scale
Change from baseline in SWN score and subitem scores | 2 weeks and 6 weeks after study treatment start
  SWN = Subjective Well-being under Neuroleptics questionnaire
Change from baseline in IMI-SR score and subitem scores | 2 weeks and 6 weeks after study treatment start
  IMI-SR = Intrinsic Motivation Inventory for Schizophrenia Research (questionnaire)
CGI-I score | 2 weeks and 6 weeks after study treatment start
  CGI-I = Clinical Global Impression if Improvement
Change from baseline in BARS total and subitem scores | 6 weeks after study treatment start
  BARS = Barnes Akathisia Rating Scale
Change from baseline in BACS score and subitem scores | 1 day, 2 weeks and 6 weeks after study treatment start
  BACS = Brief Assessment of Cognition Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marc De Hert, M.D., PhD, Principal Investigator — University Psychiatric Institute Sint-Jozef Leuvensesteenweg 517 B-3070 Kortenberg, Belgium
Locations (1):
- University Psychiatric Institute Sint-Jozef, Kortenberg, Belgium